CLINICAL TRIAL: NCT02457156
Title: PANasta Trial Cattell-Warren Versus Blumgart Techniques of Pancreatico-jejunostomy Following Pancreato-duodenectomy - a Double Blinded Multi Centred Trial
Brief Title: Cattell-Warren Versus Blumgart Techniques of Pancreatico-jejunostomy Following Pancreato-duodenectomy
Acronym: PANasta
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UoL000732
Record Dates: First submitted 2015-03-05; First posted 2015-05-29 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatico-jejunostomy; Pancreato-duodenectomy; Cattell-Warren anastomosis; Blumgart anastomosis
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blumgart Anastomosis (Experimental): Re-construction of the pancreatic remnant following pancreatico-duodenectomy using a "Blumgart" method of pancreatico-jejunostomy.
  Octreotide will be administered.
  Interventions: Procedure: Blumgart Anastomosis; Drug: Octreotide
- Cattell-Warren Anastomosis (Active Comparator): Re-construction of the pancreatic remnant following pancreato-duodenectomy using a "Cattell-Warren" method of pancreatico-jejunostomy.
  Octreotide will be administered.
  Interventions: Procedure: Cattell-Warren Anastomosis; Drug: Octreotide

INTERVENTIONS:
Procedure: Blumgart Anastomosis — 1. Trans pancreatic suture "U" stich incorporating pancreatic parenchyma and jejunal serosa, left loose.
  2. Pancreatic duct to jejunal mucosa sutures, inserted and tied.
  3. Trans pancreatic suture "U" stich brought back through the jejuanl serosa anteriorly, tied.
  Other Names: Pancreatico-jejunostomy
  Arms: Blumgart Anastomosis
Procedure: Cattell-Warren Anastomosis — 1. Posterior row of sutures from pancreatic parenchyma to jejunal serosa, inserted and tied.
  2. Pancreatic duct to jejunal mucosa sutures, inserted and tied.
  3. Anterior row of sutures from pancreatic parenchyma to jejunal serosa, inserted and tied.
  Other Names: Pancreatico-jejunostomy
  Arms: Cattell-Warren Anastomosis
Drug: Octreotide — Octrotide (100ug) to be administered on the evening before surgery and then 100ug three times daily on the day of surgery and post operative days 1 - 6.
  Other Names: Sandostatin

SUMMARY:
The purpose of this study is to compare two different techniques of performing a pancreatic anastomosis; Cattell-Warren versus Blumgart to determine if a Blumgart anastomosis reduces pancreatic remnant leak, post-operative complications and overall length of hospital stay.

DETAILED DESCRIPTION:
This is a randomised controlled, phase III, double blinded, multicentre clinical trial comparing Cattell-Warren (CWA) versus. Blumgart (BA) methods of pancreaticojejunostomy following pancreaticduodenectomy for supected malignancy of the pancreatic head.

The primary objective of the trial is to establish if the Blumgart anastomosis reduces pancreatic remnant leak and in turn complications, hospital stay, cost and promote enhanced recorvery programs.

506 patients (253 patients per treatment arm) will be recruited from approximately 7 centres throughout the United Kingdom.

Patients recommended for resection who provide written informed consent will be randomised to one of the following treatment arms on the day of surgery by the surgeon:

Arm A: Blumgart method of panreaticojejunostomy. Arm B: CattellWarren method pf pancreaticojejunostomy.

Randomisation will be undertaken intra-operatively, following pancreatic head excision, just prior to pancreatic head remnant reconstruction.

Patients will be assessed post operatively on days 3 to 7 and on day of dishcharge from hospital. Patients will continue to be followed up in the outpatient setting at 3, 6 and 12 months post surgery.

All laboratory and physical assessments performed will be in line standard care.

Blood samples for the translational study will be taken subject to informed consent pre-operatively and post-operatively 5 days after surgery.

A histological (H&E stained) slide of the pancreatic transection margin should be taken as routine. This will be requested from each patient for central pathology review to assess the amount of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective pancreato-duodenectomy for presumed malignancy.
* Ability of the subject to understand the nature and consequences of the trial.
* Ability to rovide writen informed consent.
* Age 18 or greater.

Exclusion Criteria:

* Patients undergoing extended pancreato-duodenectomy
* Left, central or total pancreatectomy.
* Arterial resection or multi-visceral resection
* Previous pancreatic surgery
* Surgery for known chronic pancreatitis.
* Recruited to any other pancreatic resection trial.
* Pregnant women.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from time of consent up to the day of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Presence or absence of post-operative pancreatic fistula | Assessed up to 3 months after surgery.
  Post-operative pancreatic fistula are defined as any abnormal connection between the pancreatic duct epithelium and another epithelised surface, which contains pancreatic derived, enzyme rich fluid. This will be assessed up to 3 months following surgery on inpatient days 3-7, day of discharge (expected to be 1 - 5 weeks after surgery) and 3 month follow up.

SECONDARY OUTCOMES:
Entry into programs of adjuvent therapy | 3, 6 and 12 month follow up
Mortality Rate | Death due to any cause during the study will be recorded
Rate of delayed gastric emptying | Post operative day 3, 5, 7, and the day of discharge, which is expected to be between 1 - 5 weeks after surgery.
Rate of wound infections | Post operative day 3, 5, 7, the day of discharge, which is expected to be between 1 - 5 weeks after surgery and 3, 6 and 12 month follow up
Rate of pulmonary infection | The day of discharge, which is expected to be between 1 - 5 weeks after surgery and 3 month follow up.
Rate of post-operative fluid collections | post operative days 3-7, the day of discharge, which is expected to be between 1 - 5 weeks after surgery and 3 month follow-up
Operation time | Day of surgery
Rate of intra and post-operative bleeding | day of surgery, post operaive day 3, 5, 7 and the day of discharge, which is expected to be between 1 - 5 weeks after surgery
Rate of re-operation | Up to 12 months after surgery
Rate of venous thrombo-embolism | Post operative day 3, 5, 7, the day of discharge, which is expected to be between 1 - 5 weeks after surgery, 3, 6 and 12 month follow up
Length of hospital stay | The day of discharge, which is expected to be between 1 - 5 weeks after surgery, 3, 6 and 12 month follow-up
Quality of Life measured by the QLQ-C30 questionnaire | Enrolment, the day of discharge, which is expected to be between 1 - 5 weeks after surgery, 3, 6 and 12 month follow-up
Health economic evaluation measured by the EQ-5D questionnaire | Enrolment, the day of discharge, which is expected to be between 1 - 5 weeks after surgery, 3, 6 and 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Halloran, Principal Investigator — University of Liverpool
Locations (1):
- Royal Liverpool University Hospital, Liverpool, Merseyside, United Kingdom